CLINICAL TRIAL: NCT00547391
Title: Recurrent Throat Infections and Tonsillectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oulu University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Diary nr 106/2007
Record Dates: First submitted 2007-10-19; First posted 2007-10-22 (Estimated); Last update posted 2012-04-19 (Estimated); Status verified 2012-02

CONDITIONS: Tonsillitis; Pharyngitis
Keywords: adults; children; tonsillectomy
MeSH Terms: conditions — Tonsillitis; Pharyngitis | interventions — Tonsillectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (No Intervention): patients on waiting list for a minimum of 5 months. These patients receive no prophylactic intervention for their recurrent pharyngitis episodes.
  Interventions: Other: no intervention
- 2 (Active Comparator): Tonsillectomy as soon as possible after randomization (within 2-3 weeks).
  Interventions: Procedure: Tonsillectomy

INTERVENTIONS:
Procedure: Tonsillectomy — Tonsillectomy under general anesthesia as a day surgery using diathermy or blunt dissection. Follow up started from the day of surgery.
  Arms: 2
Other: no intervention — No intervention (controls). Follow up started from the day of randomization.
  Arms: 1

SUMMARY:
The purpose of this study is to find out if tonsillectomy reduces the short-term risk of having an objectively confirmed (sequential changes in serum crp and procalcitonin levels) delayed pharyngitis episode among patients suffering from recurrent pharyngitis episodes. Other aims are to find out the effect of tonsillectomy to reduce the number of pharyngitis episodes or symptoms. Still, the possible disadvantages of tonsillectomy and changes in the quality of life after tonsillectomy among these patients are examined.

DETAILED DESCRIPTION:
We will have a prospective randomized study. We allocated 87 consecutive patients referred for tonsillectomy randomly in two groups: tonsilectomy group or waiting list(control group). Patients in tonsillectomy group were operated as soon as possible and data on postoperative morbidity was collected. In the control group, patients were placed on our normal waiting list and they were operated on in normal time (about 5-6 months). The data on preoperative morbidity was collected. All the pharyngitis episodes were treated by a study investigator and laboratory tests (crp, procalcitonin) were taken at that time and after three days. In addition, the patients record their symptoms on a diary.

ELIGIBILITY:
Inclusion Criteria:

* Patients selected among the cases referred to tonsillectomy for recurrent pharyngitis episodes to a tertiary care university ENT clinic (Oulu, Finland).
* At least three pharyngitis episodes difficult enough for the patients to seek for medical attention during the past 12 months

Exclusion Criteria:

* Patients with other serious diseases (day surgery not feasible)
* Patients having long time antibiotic treatment for other disease
* Patients diagnosed to have peritonsillar abscess
* Pregnancy
* Age of 12 or under
* Patients living outside Oulu or its 8 neighbouring cities (day surgery not feasible)
* Patients suffering only from halitosis or bacterial plugs of palatine tonsils

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2007-11; Primary Completion 2010-12 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Absolute percentage difference between groups of patients having pharyngitis with delayed recovery time defined by symptoms and blood sample values (crp, procalcitonin) | 5 months follow up

SECONDARY OUTCOMES:
Absolute percentage difference of patients having group A streptococcal pharyngitis. | 5 months follow up
Absolute percentage difference of patients having acute pharyngitis episode with and without medical consultation | 5 months follow up
Difference in the number and quality (mild, severe) of symptomatic days (fever, sore throat, rhinitis, cough) | 5 months follow up
Absolute percentage difference having harmful effects related to tonsillectomy (haemorrhage, soft tissue burns etc.) | 5 months follow up

CONTACTS AND LOCATIONS:
Overall Officials: Petri Koivunen, MD, Principal Investigator — Dept of Otolaryngology, University of Oulu, Finland; Aila Kristo, MD, Principal Investigator — Dept of Otolaryngology, University of Oulu, Finland; Onni Niemelä, Principal Investigator — Laboratory, University of Oulu, Finland; Markku Koskela, Principal Investigator — Microbiological Laboratory, University of Oulu, Finland; Timo J Koskenkorva, MD, Principal Investigator — Dept of Otolaryngology, University of Oulu, Finland; Olli-Pekka Alho, professor, Study Chair — Dept of Otolaryngology, University of Oulu, Finland
Locations (1):
- Oulu University Hospital, Oulu, Finland

REFERENCES:
- [Derived] Koskenkorva T, Koivunen P, Koskela M, Niemela O, Kristo A, Alho OP. Short-term outcomes of tonsillectomy in adult patients with recurrent pharyngitis: a randomized controlled trial. CMAJ. 2013 May 14;185(8):E331-6. doi: 10.1503/cmaj.121852. Epub 2013 Apr 2. PMID 23549975